CLINICAL TRIAL: NCT01967628
Title: Human Lung Responses to Respiratory Pathogens
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Alicia Gerke, Assistant Professor, University of Iowa
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: DMID 06-0003; N01AI30040-11-0-0 (NIH)
Record Dates: First submitted 2013-10-17; First posted 2013-10-23 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: Respiratory Infection
Keywords: Vitamin D; Respiratory infection; Innate immunity
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (cholecalciferol) (Experimental): Vitamin D3 (1000 international units) daily for 3 months.
  Interventions: Dietary Supplement: Vitamin D3 (cholecalciferol)
- Sugar capsule (Placebo Comparator): Placebo comparator made of sugar in a capsule
  Interventions: Dietary Supplement: Placebo Sugar Pill

INTERVENTIONS:
Dietary Supplement: Vitamin D3 (cholecalciferol)
  Arms: Vitamin D3 (cholecalciferol)
Dietary Supplement: Placebo Sugar Pill
  Arms: Sugar capsule

SUMMARY:
For most individuals, the lung has a remarkable ability to deal with exposure to a variety of inhaled bacteria. Some individuals, however, do have recurrent bacterial infections, usually in the form of acute or chronic bronchitis and, in some instances, pneumonia. The reasons for this variability in bacterial infections between otherwise healthy subjects, between types of lung disease, and within the same type of lung disease are poorly understood.

Variability in susceptibility to bacterial infections is partially explained by differences in exposure to infectious agents, genetic susceptibility and innate (or early) immune responses. It is of interest that the incidence and severity of bacterial infections is greatest during the winter months. Other than viral infections, there are few variables that change with season. Vitamin D is one known immune modulator with a seasonal periodicity. The hypothesis of this study is that levels of vitamin D are an important determinant of the innate defense of the lung against inhaled bacteria. The investigators further postulate that vitamin D has effects on the innate immune function of both alveolar macrophages and lung epithelial cells.

ELIGIBILITY:
Inclusion Criteria:

Signed informed consent form Age 18 - 60 Healthy nonsmoker, healthy smoker Forced expiratory volume in 1 second (for smokers) > 60% predicted.

Exclusion Criteria:

* Pregnant or breastfeeding
* Medications (with the exception of hormonal birth control, thyroid medication or prespecified over the counter medications), including multi-vitamins and any preparation that contains vitamin D
* Asthma
* Heart disease
* Diabetes
* Previous positive tuberculin skin test, or previous diagnosis of tuberculosis
* Recent respiratory tract infection
* History of multiple bouts of pneumonia
* Allergies to caines, atropine, or a history of adverse reaction to narcotics
* Other factors that increase the risk of bronchoscopy
* Evidence of acute bronchitis within the past 2 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 98 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alicia K Gerke, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

REFERENCES:
- [Derived] Vargas Buonfiglio LG, Cano M, Pezzulo AA, Vanegas Calderon OG, Zabner J, Gerke AK, Comellas AP. Effect of vitamin D3 on the antimicrobial activity of human airway surface liquid: preliminary results of a randomised placebo-controlled double-blind trial. BMJ Open Respir Res. 2017 Jun 4;4(1):e000211. doi: 10.1136/bmjresp-2017-000211. eCollection 2017. PMID 28883932
- [Derived] Gerke AK, Pezzulo AA, Tang F, Cavanaugh JE, Bair TB, Phillips E, Powers LS, Monick MM. Effects of vitamin D supplementation on alveolar macrophage gene expression: preliminary results of a randomized, controlled trial. Multidiscip Respir Med. 2014 Mar 26;9(1):18. doi: 10.1186/2049-6958-9-18. PMID 24669961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were included if they were 18-60 years old and able to understand and sign a consent form. All study procedures were performed at the University of Iowa Hospitals and Clinics bronchoscopy lab and clinical research unit between May 2008 and July 2010.
Pre-assignment Details: Subjects were included if they were 18-60 years.Subjects were excluded if taking a multivitamin or vitamin D supplement within the previous three months, pregnant or breastfeeding,had a vaccination within one month, significant comorbid conditions, respiratory infection, history of positive tuberculin skin test, or use of antibiotics recently.
Groups:
- Vitamin D3: Vitamin D3 (1000 IUs) daily for 3 months.
  Vitamin D3 (cholecalciferol)
- Sugar Capsule: Placebo comparator made of sugar in a capsule
  Placebo Sugar Pill
Period: Overall Study
Arm/Group | Vitamin D3 | Sugar Capsule
Started | 48 | 50
Completed | 21 | 19
Not Completed | 27 | 31
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Unable to complete bronchoscopy | 4 | 6
Not completed — Lost to Follow-up | 1 | 0
Not completed — Low protein concentration in sample | 20 | 25

BASELINE CHARACTERISTICS:
Groups:
- Vitamin D ASL: Analysis of airway surface liquid in those taking Vitamin D
- Placebo ASL: Analysis of airway surface liquid in those taking placebo.
- Total: Total of all reporting groups
Arm/Group | Vitamin D ASL | Placebo ASL | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.8 (7.6) | 29.4 (13) | 26 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 15 | 11 | 26
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 20 | 16 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smokers [Count of Participants; unit: Participants] | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Antimicrobial Activity by Airway Surface Liquid (ASL) as Measured by Relative Light Units (RLU)
Description: We investigated the effect of vitamin D3 supplementation on airway surface liquid antimicrobial activity using a bioluminescent bacterial challenge. We challenged airway surface liquid samples with bioluminescent bacteria and measured live bacteria by relative light units (RLU) after 2 minutes as a surrogate of antimicrobial activity. We interpreted a reduction in live bacteria after challenge in relative light units as increased antimicrobial activity
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: Relative Light Units (RLU)
Groups:
- Vitamin D3: Vitamin D3 (cholecalciferol) at 1000 international units daily for 3 months
Arm/Group | Vitamin D3 | Sugar Capsule
Number analyzed (Participants) | 21 | 19
Relative Light Units (RLU) | -581 [-1122 to -40] | -485 [-1170 to 199]

ADVERSE EVENTS:
Groups:
- Vitamin D Airway Surface Liquid: Analysis of airway surface liquid in those taking Vitamin D
- Placebo Airway Surface Liquid: Analysis of airway surface liquid in those taking placebo.
Arm/Group | Vitamin D Airway Surface Liquid | Placebo Airway Surface Liquid
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No